CLINICAL TRIAL: NCT05671094
Title: Implementation of a Multimodal Prehabilitation Program in Robotic Oncological Surgery: a Pilot and Feasibility Study
Brief Title: Implementation of a Multimodal Prehabilitation Program in Robotic Oncological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: f/2022/154
Record Dates: First submitted 2022-12-20; First posted 2023-01-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer; Gynecologic Cancer
Keywords: Prehabilitation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All treating physicians including surgical team, attending anesthetist and surgeon, all researcher assessing outcomes (i.e. study nurse + surgeon) and the data-managers will be blinded for group allocation until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Standard of care, i.e no specific program prior to surgery.
- Prehabilitation group (Experimental): A multimodal prehabilitation program including 4 different components (physical, cognitive, nutritional and stress reduction prehabilitation) will be proposed to patients in order for them to participate during four to two weeks pre-operatively.
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — Physical, mental, stress reducing and dietary prehabilitation programme, 4 to 2 weeks before surgery
  Arms: Prehabilitation group

SUMMARY:
Current literature on prehabilitation is broad and heterogenous. Ploussard et al initiated a multimodal one-day prehabilitation program in patients before robotic radical prostatectomy involving urology nurses, anaesthetic nurses, oncology nurse specialists, anesthesiologists, dieticians, physiotherapists etc, and observed significant improvement in terms of reduction in length of stay, blood loss, and operative time, and an increase in the proportion of ambulant surgery. Santa Mina et al observed that patients following a home-based moderate-intensity exercise prehabilitation program prior to radical prostatectomy were more fit i.e have a greater score on the 6 minutes' walk test, four weeks postoperatively compared to a control group. Regrettably, this study couldn't demonstrate a difference in length of stay or complication rate. To date, evidence for efficacy of prehabilitation in gynaecological cancer patients is limited. Several reviews and a meta-analysis indicate that the level of evidence suggesting that prehabilitation may improve postoperative outcomes is low. Moreover, there is a wide variability in applied preoperative prehabilitation programs i.e, with a uni- or multimodal approach, home-based or supervised, differences in intensity and a variety of outcomes.

Therefore, there is a need for randomized controlled trials with low risk of bias and clearly defined outcome parameters to clarify the potential benefit of prehabilitation for patients

Hence, the primary goal of this randomized pilot study is to determine the feasibility of the implementation of a multimodal prehabilitation program in patients undergoing robotic oncologic urological or gynaecological surgery in a Belgian tertiary center in terms of protocol adherence and recruitment rate.

DETAILED DESCRIPTION:
The main elements of established enhanced recovery after surgery (ERAS) include a minimally invasive surgical approach when feasible, locoregional analgesia, limited use and duration of drains, minimized blood loss and perioperative fluid administration, early oral re-nutrition, respiratory physiotherapy, and early mobilization. These pathways have demonstrated to be beneficial in the oncological surgery field by reducing hospitalization costs and peri-operative complications, while maintaining suitable oncological and functional outcomes. It has to be emphasized that patients who are active and well-functioning prior to surgery, have fewer complications, recuperate faster, and experience better recovery compared to their less fit counterparts. Recently, prehabilitation as a strategy to begin the rehabilitation process before surgery gains more interest. Although there is no single definition of prehabilitation available, this intervention aims to actively prepare patients before surgery through exercise, nutritional support, psycho-cognitive training or a combination thereof.

Current literature on prehabilitation is broad and heterogenous. Ploussard et al initiated a multimodal one-day prehabilitation program in patients before robotic radical prostatectomy involving urology nurses, anaesthetic nurses, oncology nurse specialists, anesthesiologists, dieticians, physiotherapists etc, and observed significant improvement in terms of reduction in length of stay, blood loss, and operative time, and an increase in the proportion of ambulant surgery. Santa Mina et al observed that patients following a home-based moderate-intensity exercise prehabilitation program prior to radical prostatectomy were more fit i.e have a greater score on the 6 minutes' walk test, four weeks postoperatively compared to a control group. Regrettably, this study couldn't demonstrate a difference in length of stay or complication rate. To date, evidence for efficacy of prehabilitation in gynaecological cancer patients is limited. Several reviews and a meta-analysis indicate that the level of evidence suggesting that prehabilitation may improve postoperative outcomes is low. Moreover, there is a wide variability in applied preoperative prehabilitation programs i.e, with a uni- or multimodal approach, home-based or supervised, differences in intensity and a variety of outcomes.

Therefore, there is a need for randomized controlled trials with low risk of bias and clearly defined outcome parameters to clarify the potential benefit of prehabilitation for patients Hence, the primary goal of this randomized pilot study is to determine the feasibility of the implementation of a multimodal prehabilitation program in patients undergoing robotic oncologic urological or gynaecological surgery in a Belgian tertiary center in terms of protocol adherence and recruitment rate.

Study design

This is an observer-blind, randomized controlled, superiority trial. All participants will receive standardized perioperative care according to established ERAS protocols (main elements include a minimally invasive surgical approach when feasible, locoregional analgesia, limited use and duration of drains, minimized blood loss and perioperative fluid administration, early oral re-nutrition, respiratory physiotherapy, and early mobilization).

The standard preoperative pathway includes risk assessment, medication management and perioperative blood management.

Randomization

Patients will be randomly assigned in a 1:1 ratio to either of the two study groups: an intervention group undergoing the prehabilitation program and a control group. A block randomization of 4, stratified per type of surgery, will be performed using a computer-generated random allocation sequence, created by the study statistician. Allocation numbers will be sealed in opaque envelopes, which will be opened in sequence by an unblinded member of the study team after enrollment of a patient into the study. The randomization list will remain with the study statistician for the whole duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* Competent to provide informed consent
* Undergoing robotic oncological urological or gynaecological surgery in ≥ 30 days from enrollment.
* Fluent in Dutch

Exclusion Criteria:

* Premorbid conditions or orthopedic impairments with contraindications to exercise
* Cognitive disabilities defined as evolutive neurological or neurodegenerative disease
* ASA score 4 or higher or patient under palliative care
* Expected length of stay at hospital < 48 hours
* Patient under tutorship or curatorship
* Pregnant or breast-feeding woman
* Absence of informed consent or request to not participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence rate to the prehabilitation program | throughout study completion, an average of 1 year
  Protocol adherence is defined as excellent if 80% of patients were fully adherent to the prehabilitation program. Full adherence is defined as adherence to all 4 different prehabilitation program components (see above). Adherence to the physical component will be assessed by the physical medicine and rehabilitation physician, responsible for this component. Adherence to the nutrition component will be assessed by the dietician, responsible for coaching of patients with nutrition. The other 2 components will be assessed by the study team at the end of the program.
Recruitment rate | 6 months after the start of the study
  Recruitment rate is defined as excellent if 40 patients can be enrolled in this study in a time frame of 6 months.

SECONDARY OUTCOMES:
Incidence of Postoperative Cognitive Disorder | 3 months after surgery
  A battery of four tests (Rey Auditory Verbal Learning Test (RAVLT), Trial Making Test (TMT A and B) and the Grooved Pegboard Test) mentioned by the 'statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery', published in 1995 supplemented with two additional tests (ie, the Welscher Adult Intelligence Scale (WAIS)-III digit span test and WAIS-III digit symbol-coding test) will be administered to determine the cognitive outcome. LPOCD is defined as an RCI (Reliable Change Index) ≤-1.645 (significance level 5%) or Z-score ≤-1.645 in at least two different tests.
Assessment of Patient Recovery | Baseline (before surgery) and 6 weeks after surgery.
  This will be assessed with the WHO Disability Assessment Schedule 2.0 (WHODAS) questionnaire.
Assessment of quality of recovery | Baseline (before surgery) and 24 hours after surgery
  Quality of recovery will be assessed through the QoR-40 questionnaire.
Hospital length of stay | through study completion, an average of 3 months
  Data regarding hospital admission and discharge will be collected.
Assessment of amount of red blood cell transfusion | throughout study completion, an average of 3 months
  Assessment of amount of red blood cell transfusion during the surgery and the stay in hospital.
Assessment of re-admission | through study completion, an average of 3 months
  Evaluation regarding re-admission during 3 months post-operatively will be collected
Complications | through study completion, an average of 3 months
  Assessment of complications
the 6 minutes walking test (Physical fitness) | Baseline (before surgery) and 6 weeks after surgery
  Assessment of physical fitness with the 6 minutes walking test
Physical fitness | Baseline (before surgery) and 6 weeks after surgery
  Assessment of physical fitness with the timed up and go test

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No